CLINICAL TRIAL: NCT00471965
Title: Oxaliplatin(Eloxatin®) + 5-FU/LV (FOLFOX4) Compared With Single Agent Doxorubicin (Adriamycin®) as Palliative Chemotherapy in Advanced Hepatocellular Carcinoma Patients Ineligible for Curative Resection or Local Treatment
Brief Title: Oxaliplatin + 5-FluoroUracil/LeucoVorin (5-FU/LV) (FOLFOX4) Versus Doxorubicin as Palliative Chemotherapy in Advanced Hepatocellular Carcinoma Patients
Acronym: EACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXALI_L_00858
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Oxaliplatin + 5-Fluorouracil/Leucovorin
  Interventions: Drug: Oxaliplatin + 5-Fluorouracil/Leucovorin
- B (Active Comparator): Doxorubicin
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Oxaliplatin + 5-Fluorouracil/Leucovorin — Day 1: Oxaliplatin 85mg/m² 2h IV infusion, leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m2 22h IV infusion.
  Day 2: Leucovorin 200mg/m² 2h IV infusion, 5-fluorouracil 400mg/m² IV bolus, 5-fluorouracil 600mg/m² 22h IV infusion.
  Repeated every 2 weeks
  Arms: A
Drug: Doxorubicin — Day 1: Doxorubicin 50mg/m² iv infusion. Repeated every 3 weeks.
  Arms: B

SUMMARY:
Primary:

* Overall Survival (OS)

Secondary:

* Time to Tumor Progression (TTP)
* Response Rate (RR)
* Improvement of Quality of Life (QoL)
* Safety
* Secondary resection rate

ELIGIBILITY:
Inclusion Criteria:

* Histologically, cytologically or clinically diagnosed (in patient with cirrhosis, Alpha-Fetoprotein(AFP)≥400μg/L and morphological evidence [contrast Computed Tomography(CT)/Magnetic Resonance Imaging(MRI)] of hypervascular liver tumor, elevated AFP level due to other reasons [germ cell carcinoma, progressive chronic hepatitis, pregnancy, etc] can be excluded) unresectable hepatocellular carcinoma, ineligible or if the patient does not consent to receive local invasive treatment (chemo-embolism, ablation, etc.).
* At least one measurable lesion (on CT: ≥2cm, on spiral CT or MRI ≥1cm)
* Have not received previous palliative systemic chemotherapy for metastatic disease. If the patient received previous systemic chemotherapy as adjuvant treatment, he must have been completed at least 12 months previously.
* Patients progress after previous local treatment and at the time of randomization is at least 4 weeks after the last interventional therapy (Hepatic Artery Infusion, Trans-Artery Embolization or Trans-Artery Chemo-Embolization) or at least 8 weeks after the last radiotherapy/ablation/ Percutaneous Ethanol Injection to the target lesion.
* Karnofsky Performance Score≥70, Barcelona of Cancer Liver Category stage B/C
* Patients must have adequate organ and marrow function:

  * Neutrophilus≥1.5X10^9/L
  * Platelets≥75X10^9/L
  * Asparagine AminoTransferase,Alanine AminoTransferase<2.5 Upper Normal Limit(UNL)
  * Total Bilirubin<1.5 UNL
  * International Normalized Ratio<1.5
  * Child stage A or B
  * Normal base line Left Ventricular Ejection Fraction (LVEF result must be above or equal to the lower limit of normal for the institution)

Exclusion Criteria:

* Documented allergy to platinum compound or to other study drugs.
* Any previous oxaliplatin or doxorubicin treatment, except adjuvant treatment more than 12 months before the randomization.
* Previous liver transplantation.
* Patients concomitantly receiving any other anti-cancer therapy, including interferon-α and herbal medicine which was approved by local authority to be used as "anti-cancer" medicine, except radiotherapy to non-target lesion (bone metastasis, etc)
* Patients who are receiving any other study treatments.
* Pregnant or lactating women or women of childbearing potential without proper contraceptive methods.
* History of other malignant diseases, except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* Central nervous system metastasis
* Other serious illness or medical conditions

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization to the date of death due to any cause

SECONDARY OUTCOMES:
Time to progression | From the date of randomization to documentation of progression
Response rate, secondary resection rate, quality of life | From the date of randomization to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Blayney, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis Administrative Office, Shanghai, China
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand

REFERENCES:
- [Derived] Qin S, Cheng Y, Liang J, Shen L, Bai Y, Li J, Fan J, Liang L, Zhang Y, Wu G, Rau KM, Yang TS, Jian Z, Liang H, Sun Y. Efficacy and safety of the FOLFOX4 regimen versus doxorubicin in Chinese patients with advanced hepatocellular carcinoma: a subgroup analysis of the EACH study. Oncologist. 2014 Nov;19(11):1169-78. doi: 10.1634/theoncologist.2014-0190. Epub 2014 Sep 15. PMID 25223462